CLINICAL TRIAL: NCT00710983
Title: Investigating the Mortality and the Morbidity Impact of Oral Polio Vaccine at Birth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Responsible Party: Peter Aaby, Bandim Health Project
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-7041-122
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Infant, Newborn; Healthy
Keywords: Mortality; Morbidity; Growth; Immunology
MeSH Terms: interventions — Poliovirus Vaccine, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Oral polio vaccine
  Interventions: Biological: Oral polio vaccine
- B (No Intervention): No oral polio vaccine

INTERVENTIONS:
Biological: Oral polio vaccine
  Arms: A

SUMMARY:
Our group has discovered that routine vaccinations in childhood may have non-specific and sex-differential effects on overall mortality. The effects are so large that they may have marked effects on overall mortality and seriously distort female-to-male mortality rates in high-mortality settings. We recently experienced periods during which oral polio vaccine (OPV) was lacking. Hence, some children did not get the recommended OPV at birth. We were following all infants as a part of a vitamin A supplementation trial. Surprisingly, we discovered that not receiving OPV was associated with significantly lower mortality in boys, but not in girls. We bled a subgroup of the children. Receiving OPV at birth significantly dampened the immunological response to BCG given at birth in both sexes. Based on these observations, receiving OPV at birth may have two negative effects, first, it may increase male mortality, and second, it may interfere with immunity against tuberculosis. OPV at birth is given for logistic reasons, to boost polio immunity. There have been no polio cases in Guinea-Bissau for the last 10 years. Hence, there is every reason to test in a randomised trial whether not receiving OPV at birth is associated with 1) mortality, morbidity and growth and 2) immunological response to BCG.

ELIGIBILITY:
Inclusion Criteria:Normal birth weight, no overt illness or gross malformations -

Exclusion Criteria:

-

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2008-07; Primary Completion 2014-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Mortality by sex

SECONDARY OUTCOMES:
Morbidity, growth, immunology

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Derived] Lund N, Andersen A, Hansen AS, Jepsen FS, Barbosa A, Biering-Sorensen S, Rodrigues A, Ravn H, Aaby P, Benn CS. The Effect of Oral Polio Vaccine at Birth on Infant Mortality: A Randomized Trial. Clin Infect Dis. 2015 Nov 15;61(10):1504-11. doi: 10.1093/cid/civ617. Epub 2015 Jul 28. PMID 26219694
- [Derived] Eriksen HB, Biering-Sorensen S, Lund N, Correia C, Rodrigues A, Andersen A, Ravn H, Aaby P, Jeppesen DL, Benn CS. Factors associated with thymic size at birth among low and normal birth-weight infants. J Pediatr. 2014 Oct;165(4):713-21. doi: 10.1016/j.jpeds.2014.06.051. Epub 2014 Jul 30. PMID 25085521